CLINICAL TRIAL: NCT03504917
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Efficacy, and Safety Study of Balovaptan in Adults With Autism Spectrum Disorder With a 2-Year Open-Label Extension
Brief Title: A Study of Balovaptan in Adults With Autism Spectrum Disorder With a 2-Year Open-Label Extension
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A futility analysis assessed that the study is highly unlikely to meet the pre-defined primary objective of the study. No new safety concerns were identified.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN39434
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — balovaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Balovaptan (Experimental)
  Interventions: Drug: Balovaptan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Balovaptan — Participants will receive 10 mg of oral administration balovaptan once a day (QD).
  Arms: Balovaptan
Drug: Placebo — Participants will receive matching placebo.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of 10 mg of oral administration balovaptan once a day (QD) compared with matching placebo in adults (18 years and older) with autism spectrum disorder (ASD).

ELIGIBILITY:
Inclusion Criteria:

* Subject meets the DSM-5 criteria for ASD for an autism diagnosis and is confirmed using ADOS-2 criteria
* SRS-2, proxy version, total t-score >=66 at screening
* A full scale IQ score >=70 on the WASI®-II
* Subject has an appropriate study partner, in the opinion of the investigator
* For women of childbearing potential: agreement to remain abstinent or use a contraceptive method with a failure rate of <1% per year during the treatment period and for at least 28 days after the last dose of study drug
* Treatment with permitted medications (at a stable dose for 12 weeks before screening) and behavioral therapy regimens (regimens stable for 6 weeks before screening), with the intent that such treatments remain stable throughout the study and with no expected changes before the Week 24 visit

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention to become pregnant during the study
* Previous initiation of new or major change in psychosocial intervention within 6 weeks prior to screening
* Unstable or uncontrolled clinically significant affective or psychotic disorders and/or neurologic disorder that may interfere with the assessment of safety or efficacy endpoints
* Substance use disorders during the last 12 months
* Significant risk for suicidal behavior, in the opinion of the investigator
* Epilepsy or seizure disorder considered not well controlled within the past 6 months or changes in anticonvulsive therapy within the last 6 months
* Clinical diagnosis of peripheral neuropathy
* Within the last 2 years, unstable or clinically significant cardiovascular disease
* Uncontrolled hypertension
* Unexplained syncopal episode within the last 12 months
* Confirmed elevation above upper limit of normal of CK-MB, high sensitivity cardiac troponin T, cardiac troponin I, and/or N-terminal pro B-type natriuretic peptide
* Positive serology results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) 1 or 2
* History of coagulopathies, bleeding disorders, blood dyscrasias, hematological malignancies, myelosuppression (including iatrogenic), or current major bleeding event
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or what would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Confirmed clinically significant abnormality in parameters of hematology
* Confirmed clinically significant abnormality in parameters of clinical chemistry, coagulation, or urinalysis
* Medical history of malignancy, if not considered cured

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (51):
- United States (32):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - University of California , Los Angeles (UCLA); Child, Adolescent Psychiatry, Los Angeles, California
  - PCSD Feighner Research, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Yale University / Yale-New Haven Hospital, New Haven, Connecticut
  - Sarkis Clinical Trials, Gainesville, Florida
  - APG- Advanced Psychiatric Group, Orlando, Florida
  - IMIC Inc., Palmetto Bay, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Uni of Chicago; Centre For Advanced Medicine, Chicago, Illinois
  - Lake Charles Clinical Trials, LLC, Lake Charles, Louisiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Millennium Psychiatric Associates, LLC, St Louis, Missouri
  - Hapworth Research Inc., New York, New York
  - Center for Autism and the Developing Brain, New York, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - University Hospitals, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - UPMC Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center; Department of Psychiatry, Nashville, Tennessee
  - BioBehavioral Research of Austin, PC, Austin, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Aspen Clinical Research, Orem, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Children's Hospital, Seattle, Washington
- Canada (4):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Holland Bloorview Kids Rehabilitation Hospital; Autism Research Centre, East York, Ontario
  - University of Western Ontario, London, Ontario
  - McGill University Health Centre - Glen Site, Montreal, Quebec
- France (3):
  - Hopital Charles Perrens; Centre de Ressources Autisme Aquitaine, Bordeaux
  - Hospices Civils de Lyon; Centre d'Investigation Clinique Pédiatrique, Lyon
  - Centre hospitalier du Rouvray; CRAHN Centre de Ressources Autisme Haute-Normandie, Sotteville-lès-Rouen
- Italy (4):
  - ASST di Pavia; Dip. di Scienze del Sistema Nervoso e del Comportamento, Pavia, Lombardy
  - AUSL di Piacenza; Psichiatria di Collegamento, Piacenza, Lombardy
  - ASL TO2; Centro Pilota Regione Piemonte - Dip. Salute Mentale, Turin, Piedmont
  - A.O.U. Policlinico - V. Emanuele - P.O. Gaspare Rodolico; Dip. Terapia integrata disturbi resistenti, Catania, Sicily
- Spain (4):
  - Hospital Mutua de Terrassa; Departamento de Psiquiatria, Terrassa, Barcelona
  - Hospital Universitari Vall d'Hebron; Sevicio de Psiquiatría, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Psiquiatria del niño y del adolescente, Madrid
  - Hospital Universitario Rio Hortega; Departamento de Psiquiatria, Valladolid
- United Kingdom (4):
  - Western General Hospital; Wellcome Trust CRF, Edinburgh
  - Queen Elizabeth University Hospital; Clinical Research Facility, Glasgow
  - Kings College Hospital; Kings Clinical Research Facility, London
  - RE:Cognition Health; RE:Cognition Health, London

REFERENCES:
- [Derived] Aponte EA, Tillmann J, Gleissl T, Del Valle Rubido M, Murtagh L, Sanders K, Chatham CH, Wiese T, Suter EE. Anxiety, repetitive and restricted behaviors and interests, and social communication in autistic adults: an exploratory analysis of a phase 3, randomized clinical trial. Sci Rep. 2025 Nov 6;15(1):38912. doi: 10.1038/s41598-025-22659-y. PMID 41198718
- [Derived] Jacob S, Veenstra-VanderWeele J, Murphy D, McCracken J, Smith J, Sanders K, Meyenberg C, Wiese T, Deol-Bhullar G, Wandel C, Ashford E, Anagnostou E. Efficacy and safety of balovaptan for socialisation and communication difficulties in autistic adults in North America and Europe: a phase 3, randomised, placebo-controlled trial. Lancet Psychiatry. 2022 Mar;9(3):199-210. doi: 10.1016/S2215-0366(21)00429-6. Epub 2022 Feb 10. PMID 35151410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 322 Participants were randomized. 1 Participants did not receive the treatment and in the ITT Population, 321 participants received at least one dose of the study treatment.
  The Study was discontinued early before the planned sample size was reached.
Pre-assignment Details: Participants received matching placebo in Blinded Treatment Period for 24 Weeks and 10 mg of oral administration balovaptan once a day (QD) during the Open Label Extension Treatment Period.
Groups:
- Balovaptan: Participants received 10 mg of oral administration balovaptan once a day (QD).
- Placebo: Participants received matching placebo in Blinded Treatment Period and 10 mg of oral administration balovaptan once a day (QD) in OLE Treatment period
Period: Blinded Treatment Period
Arm/Group | Balovaptan | Placebo
Started (ITT Population) | 163 | 158
Completed (ITT Population) | 103 | 102
Not Completed | 60 | 56
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 12 | 9
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 1 | 4
Not completed — Adverse Event | 4 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Unable due to leaving the study site, non-interest, withdrawal, and a partner inability | 1 | 3
Not completed — Study terminated by sponsor | 39 | 34
Not completed — Non-compliance with study drug | 0 | 1
Period: Open Label Extension Treatment Period
Arm/Group | Balovaptan | Placebo
Started (ITT Population, 63 and 61 Participants did not continue in open-label extension in Balovaptan and Placebo Arms respectively.) | 100 | 97
Completed (ITT Population) | 0 | 0
Not Completed | 100 | 97
Not completed — The participant left the study site | 0 | 1
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Lost to Follow-up | 1 | 4
Not completed — Lack of Efficacy | 3 | 1
Not completed — Adverse Event | 7 | 0
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Study terminated by sponsor | 81 | 88

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received matching placebo.
- Total: Total of all reporting groups
Arm/Group | Balovaptan | Placebo | Total
Number analyzed (Participants) | 163 | 158 | 321
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.6 (9.7) | 27.6 (9.8) | 27.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 30 | 65
  Male | 128 | 128 | 256
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 13 | 28
  Not Hispanic or Latino | 145 | 142 | 287
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 143 | 140 | 283
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 24 on the Vineland Adaptive Behavior Scales (Vineland-II) Two-domain Composite (2DC) Score.
Description: Vineland™-II Adaptive Behavior Scales 2-Domain Composite (2DC) Score is defined as mean of the Communication domain standard score & Socialization domain standard score. If any of the 2 individual domain standard scores is missing 2DC score is not computed. Vineland™-II is an instrument that measures communication, daily living skills, socialization, motor skills and maladaptive behavior of individuals with developmental disabilities. Survey Interview Form will be administered to a subject's reliable study partner in this study, during which the rater or clinician will ask to the study partner open ended questions relating to the subject's activities and behavior. Standardized scores on the Adaptive behavior composite range from 20-160 with higher scores indicating better functioning.
Time Frame: Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Balovaptan | Placebo
Number analyzed (Participants) | 111 | 99
Score | 4.56 (10.85) | 6.83 (12.18)

2. Secondary Outcome: Change From Baseline at Week 12 on the Vineland-II 2DC Score
Description: as for outcome 1
Time Frame: Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Balovaptan | Placebo
Number analyzed (Participants) | 150 | 140
Score | 3.47 (10.00) | 4.85 (12.64)

3. Secondary Outcome: Change From Baseline at Weeks 12 and 24 in the Pediatric Quality of Life (PedsQL) Inventory Generic Core Scales, Version 4.0, on Summary and Total Scores
Description: The Pediatric Quality of Life Inventory PedsQL™4.0 Generic Core Scale assessment consists of a 23 item questionnaire encompassing 4 core scale domains: Physical Functioning (8 items); Emotional Functioning (5 items); Social Functioning (5 items); and School Functioning (5 items). Items are scored on a 5 point Likert-type response scale (0=never a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; and 4=almost always a problem). Once scored, items will be reverse scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0), so that higher scores indicate better health-related quality of life.
Time Frame: Weeks 12 and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Balovaptan | Placebo
Number analyzed (Participants) | 163 | 158
Score
  Total Score at Week 12: number analyzed (Participants) | 144 | 124
  Total Score at Week 12 | 4.1 (11.2) | 5.0 (10.2)
  Psychosocial Health Summary Score at Week 12: number analyzed (Participants) | 144 | 124
  Psychosocial Health Summary Score at Week 12 | 4.9 (13.2) | 5.5 (12.7)
  Physical Health Summary Score at Week 12: number analyzed (Participants) | 144 | 125
  Physical Health Summary Score at Week 12 | 2.5 (13.3) | 4.3 (12.3)
  Total Score at Week 24: number analyzed (Participants) | 106 | 92
  Total Score at Week 24 | 8.0 (13.7) | 6.0 (11.6)
  Psychosocial Health Summary Score at Week 24: number analyzed (Participants) | 106 | 92
  Psychosocial Health Summary Score at Week 24 | 10.0 (15.4) | 6.9 (14.1)
  Physical Health Summary Score at Week 24: number analyzed (Participants) | 106 | 92
  Physical Health Summary Score at Week 24 | 4.3 (15.5) | 4.4 (14.5)

4. Secondary Outcome: Change From Baseline at Weeks 12 and 24 in the Vineland-II Adaptive Behavior Composite Standard Score
Description: The Vineland-II is an instrument that measures communication, daily living skills, socialization, motor skills (only in children up to 6 years) and maladaptive (not assessed in this study) behavior of individuals with developmental disabilities. The Survey Interview Form (i.e., semi -structured interview) will be administered to a subject's reliable study partner in this study, during which the rater or clinician will ask to the study partner open ended questions relating to the subject's activities and behavior. Domain scores will be obtained for the individual domains of Socialization, Communication, Daily Living Skills, and motor skills (up to 6 years only) and used to calculate the Vineland-II Adaptive Behavior Composite score. Standardized scores on the Adaptive behavior composite range from 20-160 with higher scores indicating better functioning. Only descriptive statistics presented instead of the planned estimated due to the early discontinuation of the study due to futility.
Time Frame: Weeks 12 and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Balovaptan | Placebo
Number analyzed (Participants) | 163 | 157
Score
  Week 12: number analyzed (Participants) | 150 | 140
  Week 12 | 2.87 (6.99) | 3.99 (10.01)
  Week 24: number analyzed (Participants) | 111 | 99
  Week 24 | 4.32 (8.43) | 5.26 (9.69)

5. Secondary Outcome: Change From Baseline at Week 12 and 24 on the Vineland-II Socialization Domain Standard Score
Description: The Vineland-II is an instrument that measures communication, daily living skills, socialization, motor skills (only in children up to 6 years) and maladaptive (not assessed in this study) behavior of individuals with developmental disabilities. The Survey Interview Form (i.e., semi -structured interview) will be administered to a subject's reliable study partner in this study, during which the rater or clinician will ask to the study partner open ended questions relating to the subject's activities and behavior. Domain scores will be obtained for the individual domains of Socialization, Communication, Daily Living Skills, and motor skills (up to 6 years only) and used to calculate the Vineland-II Adaptive Behavior Composite score. Standardized scores on the Adaptive behavior composite range from 20-160 with higher scores indicating better functioning.
  Only descriptive statistics presented instead of the planned estimand due to the early discontinuation of the study due to futility.
Time Frame: Baseline, Weeks 12 and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Balovaptan | Placebo
Number analyzed (Participants) | 163 | 158
Score
  12 Week: number analyzed (Participants) | 150 | 140
  12 Week | 3.63 (11.58) | 5.26 (12.71)
  24 Week: number analyzed (Participants) | 111 | 99
  24 Week | 5.54 (13.54) | 6.86 (11.75)

6. Secondary Outcome: Change From Baseline at Weeks 12 and 24 on the Vineland-II Communication Domain Standard Score
Description: The Vineland-II is an instrument that measures communication, daily living skills, socialization, motor skills (only in children up to 6 years) and maladaptive (not assessed in this study) behavior of individuals with developmental disabilities. The Survey Interview Form (i.e., semi -structured interview) will be administered to a subject's reliable study partner in this study, during which the rater or clinician will ask to the study partner open ended questions relating to the subject's activities and behavior. Domain scores will be obtained for the individual domains of Socialization, Communication, Daily Living Skills, and motor skills (up to 6 years only) and used to calculate the Vineland-II Adaptive Behavior Composite score. Standardized scores on the Adaptive behavior composite range from 20-160 with higher scores indicating better functioning.
Time Frame: Weeks 12 and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Balovaptan | Placebo
Number analyzed (Participants) | 163 | 158
Score
  Week 12: number analyzed (Participants) | 150 | 140
  Week 12 | 3.30 (13.74) | 4.44 (16.58)
  Week 24: number analyzed (Participants) | 111 | 99
  Week 24 | 3.59 (16.30) | 6.81 (17.50)

7. Secondary Outcome: Change From Baseline at Weeks 12 and 24 on the Vineland-II Daily Living Skills Domain Standard Score
Description: as for outcome 4
Time Frame: Weeks 12 and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Balovaptan | Placebo
Number analyzed (Participants) | 163 | 158
Score
  Week 12: number analyzed (Participants) | 150 | 140
  Week 12 | 2.93 (8.44) | 2.74 (9.20)
  Week 24: number analyzed (Participants) | 111 | 99
  Week 24 | 5.14 (9.34) | 3.02 (9.04)

8. Secondary Outcome: Change From Baseline in Severity of Clinical Impressions as Measured by Clinical Global Impression-Severity (CGI-S)
Description: The CGI-S reflects the rater's impression of the subject's current autism severity on a 7-point scale ranging from no symptoms (1) to very severe symptoms (7). Changes in CGI-S score were calculated as increase or decrease in absolute CGI-S scores between Baseline and Weeks 12 and 24. Percentage of participants reported for each change in score from baseline.
Time Frame: Weeks 12 and 24
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Balovaptan | Placebo
Number analyzed (Participants) | 147 | 136
Percentage of Participants
  Week 12 -3 | 0 | 0
  Week 12 -2 | 2.0 | 2.2
  Week 12 -1 | 21.8 | 25.0
  Week 12 0 | 74.8 | 72.1
  Week 12 +1 | 0.7 | 0.7
  Week 12 +2 | 0.7 | 0
  Week 12 +3 | 0 | 0
  Week 24 -3: number analyzed (Participants) | 109 | 100
  Week 24 -3 | 0 | 1.0
  Week 24 -2: number analyzed (Participants) | 109 | 100
  Week 24 -2 | 5.5 | 10.0
  Week 24 -1: number analyzed (Participants) | 109 | 100
  Week 24 -1 | 27.5 | 20.0
  Week 24 0: number analyzed (Participants) | 109 | 100
  Week 24 0 | 66.1 | 68.0
  Week 24 +1: number analyzed (Participants) | 109 | 100
  Week 24 +1 | 0.9 | 1.0
  Week 24 +2: number analyzed (Participants) | 109 | 100
  Week 24 +2 | 0 | 0
  Week 24 +3: number analyzed (Participants) | 109 | 100
  Week 24 +3 | 0 | 0

9. Secondary Outcome: Improvements in Clinical Impressions, as Measured by Clinical Global Impression-Improvement (CGI-I)
Description: This is a 7-point Likert scale that assesses improvement of the patient's condition. Scores range from the worst score of 7 (Very much worse) to the best score of 1 (Very much improved). Lower scores are better on this scale, and indicate greater improvement. Percentage of participants reported for each score.
Time Frame: Weeks 12 and 24
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Balovaptan | Placebo
Number analyzed (Participants) | 148 | 136
Percentage of Participants
  Week 12 1 | 0 | 0
  Week 12 2 | 10.1 | 14.7
  Week 12 3 | 36.5 | 43.4
  Week 12 4 | 50.0 | 41.2
  Week 12 5 | 3.4 | 0.7
  Week 12 6 | 0 | 0
  Week 12 7 | 0 | 0
  Week 24 1: number analyzed (Participants) | 109 | 100
  Week 24 1 | 0 | 2.0
  Week 24 2: number analyzed (Participants) | 109 | 100
  Week 24 2 | 15.6 | 24.0
  Week 24 3: number analyzed (Participants) | 109 | 100
  Week 24 3 | 44.0 | 40.0
  Week 24 4: number analyzed (Participants) | 109 | 100
  Week 24 4 | 38.5 | 33.0
  Week 24 5: number analyzed (Participants) | 109 | 100
  Week 24 5 | 0.9 | 1.0
  Week 24 6: number analyzed (Participants) | 109 | 100
  Week 24 6 | 0.9 | 0
  Week 24 7: number analyzed (Participants) | 109 | 100
  Week 24 7 | 0 | 0

10. Secondary Outcome: Change From Baseline at Weeks 12 and 24 in the Hamilton Anxiety Rating Scale (HAM-A) Total and Domain Scores
Description: The HAM-A is a 14-item, rater administered interview, assessing the severity of anxiety symptoms during the past 7 days. Seven items assess psychic anxiety and seven assess somatic anxiety. Each item utilizes a 5-point symptom severity response scale, ranging from none (0) to very severe (4). A total score is calculated that ranges from 0 to 56; higher scores are indicative of more severe anxiety.
Time Frame: Weeks 12 and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Balovaptan | Placebo
Number analyzed (Participants) | 163 | 158
Score
  Week 12 Total: number analyzed (Participants) | 153 | 143
  Week 12 Total | -1.7 (4.9) | -2.8 (4.4)
  Week 12 Psychic Anxiety Subscale: number analyzed (Participants) | 153 | 143
  Week 12 Psychic Anxiety Subscale | -1.3 (3.5) | -1.8 (3.2)
  Week 12 Somatic Anxiety Subscale: number analyzed (Participants) | 153 | 143
  Week 12 Somatic Anxiety Subscale | -0.4 (2.4) | -1.0 (2.5)
  Week 24 Total: number analyzed (Participants) | 115 | 104
  Week 24 Total | -2.7 (4.5) | -2.8 (5.7)
  Week 24 Psychic Anxiety Subscale: number analyzed (Participants) | 115 | 104
  Week 24 Psychic Anxiety Subscale | -2.1 (3.4) | -1.8 (3.9)
  Week 24 Somatic Anxiety Subscale: number analyzed (Participants) | 115 | 104
  Week 24 Somatic Anxiety Subscale | -0.6 (2.2) | -0.1 (2.9)

11. Secondary Outcome: Proportion of Subjects With a >=6-point Improvement in Vineland-II 2DC Score
Description: The Vineland-II is an instrument that measures communication, daily living skills, socialization, motor skills (only in children up to 6 years) and maladaptive (not assessed in this study) behavior of individuals with developmental disabilities. The Survey Interview Form (i.e., semi -structured interview) will be administered to a subject's reliable study partner in this study, during which the rater or clinician will ask to the study partner open ended questions relating to the subject's activities and behavior. Domain scores will be obtained for the individual domains of Socialization, Communication, Daily Living Skills, and motor skills (up to 6 years only) and used to calculate the Vineland-II Adaptive Behavior Composite score. Standardized scores on the Adaptive behavior composite range from 20-160 with higher scores indicating better functioning
  All participants who have an improvement of at least 6 points are included in the >=6 score threshold
Time Frame: Weeks 12 and 24
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Balovaptan | Placebo
Number analyzed (Participants) | 128 | 114
Percentage of Participants
  Week 12 >=6 | 34.4 | 42.1
  Week 24 >=6: number analyzed (Participants) | 100 | 93
  Week 24 >=6 | 43 | 48.4

12. Secondary Outcome: Percentage of Participants With Adverse Events
Description: According to the ICH guideline for Good Clinical Practice, an adverse event is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution.
  The Blinded Treatment Period continued for 24 weeks, Open Label Extension (OLE) Treatment Period continued up to 2 years. The study was pre-maturely terminated, therefore did not reach the planned end date.
Time Frame: Week 24 and Up to Approximately 2 Years
Population: Safety Population
Measure: Number; unit: Percentage of Participants
Groups:
- Balovaptan Treatment: Participants received 10 mg of oral administration balovaptan once a day (QD). Blinded Treatment Period
- Placebo Treatment: Participants received matching placebo. Blinded Treatment Period
- Balovaptan OLE: Participants received 10 mg of oral administration balovaptan once a day (QD). OLE Treatment Period
- Placebo OLE: Participants received matching placebo in Blinded Treatment Period and 10 mg of oral administration balovaptan once a day (QD). OLE Treatment Period
Arm/Group | Balovaptan Treatment | Placebo Treatment | Balovaptan OLE | Placebo OLE
Number analyzed (Participants) | 163 | 158 | 100 | 97
Percentage of Participants | 60.1 | 65.8 | 59.0 | 55.7

ADVERSE EVENTS:
Time Frame: From baseline to the end of Safety Period, up to 2 years
Description: The proportion of patients with at least one AE in the balovaptan and placebo treatment arms in the Blinded Treatment period and Open Label Extension (OLE)Treatment period.
  Other Adverse Events are reported at 5% frequency threshold. In the Open Label Extension (OLE) Treatment Period, the participants received active treatment, i.e. 10mg balovaptan QD. Placebo was only given during the blinded treatment period but not during OLE Treatment Period.
Groups:
- Balovaptan in Blinded Treatment Period; Balovaptan in Open Label Extension Treatment Period: Participants received 10 mg of oral administration balovaptan once a day (QD).
- Placebo Blinded Treatment Period: Participants received matching placebo.
- Placebo in Open Label Extension Treatment Period: Participants received matching placebo in Blinded Treatment Period and 10 mg of oral administration balovaptan once a day (QD). OLE Treatment Period
Arm/Group | Balovaptan in Blinded Treatment Period | Placebo Blinded Treatment Period | Balovaptan in Open Label Extension Treatment Period | Placebo in Open Label Extension Treatment Period
All-Cause Mortality (participants affected / at risk) | 0/163 | 1/158 | 0/100 | 0/97
Serious Adverse Events (participants affected / at risk) | 2/163 | 5/158 | 0/100 | 2/97
Other Adverse Events (participants affected / at risk) | 49/163 | 59/158 | 28/100 | 30/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balovaptan in Blinded Treatment Period (N=163) | Placebo Blinded Treatment Period (N=158) | Balovaptan in Open Label Extension Treatment Period (N=100) | Placebo in Open Label Extension Treatment Period (N=97)
Panic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balovaptan in Blinded Treatment Period (N=163) | Placebo Blinded Treatment Period (N=158) | Balovaptan in Open Label Extension Treatment Period (N=100) | Placebo in Open Label Extension Treatment Period (N=97)
Diarrhoea (Gastrointestinal disorders) | 11 (15) | 14 (15) | 5 (5) | 4 (4)
Nasopharyngitis (Infections and infestations) | 14 (14) | 19 (22) | 7 (10) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 10 (13) | 9 (11) | 6 (7) | 7 (11)
Dizziness (Nervous system disorders) | 2 (2) | 10 (10) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 8 (13) | 7 (9) | 5 (5) | 10 (17)
Anxiety (Psychiatric disorders) | 8 (11) | 7 (7) | 8 (8) | 3 (4)
Insomnia (Psychiatric disorders) | 5 (5) | 8 (8) | 3 (3) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (8) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (8) | 1 (1) | 5 (5)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT03504917/Prot_SAP_000.pdf